CLINICAL TRIAL: NCT04237311
Title: Effect and Mechanism of Bariatric Surgery on Male Reproductive Function
Brief Title: Bariatric Surgery and Male Reproductive Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 20191107
Record Dates: First submitted 2019-12-25; First posted 2020-01-23 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Bariatric Surgery Candidate; Roux en Y Gastric Bypass; Sleeve Gastrectomy
Keywords: Semen; Micronutrient; Inflammation; Nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Inflammation | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic sleeve gastrectomy is performed as following: after greater curvature dissociating, the gastric tube was calibrated over a 36F bougie and transection started approximately 5-6 cm from the pylorus toward the left diaphragmatic crus, using linear cutting stapler of 3.5- or 4.8-mm-high staples, depending on gastric thickness.
Procedure: Roux-en-Y gastric bypass — Laparoscopic Roux-en-Y gastric bypass is performed as following: a gastric pouch of approximately 30mL was obtained using linear cutting stapler, the sum of the length of the alimentary limb and the biliopancreatic limb> 200 cm (can be adjusted according to the incidence of the patient's BMI, type 2 diabetes mellitus and the specific situation).

SUMMARY:
Obesity is a global public health problem. According to literature reports, as of 2016, China's obese population has reached more than 90 million and type 2 diabetes mellitus has reached more than 100 million, which has brought a serious health and economic burden to China. In addition to various health problems such as cardiovascular, osteoarthritis, and tumors, obesity can also cause abnormalities in reproductive endocrine. In women, it can cause abnormal menstruation, polycystic ovary syndrome, and male obesity can cause secondary gonadal. Hypofunction (MOSH). MOSH is an endocrine dysfunction. It is reported to have a prevalence of approximately 45% in moderate to severe obesity. In addition, studies have pointed out that the prevalence of hypogonadism in men with type 2 diabetes and obesity higher. However, there are no studies on the reproductive function of Chinese male patients after bariatric surgery. Pre- and post-operative semen will be collected for analysis to observe the effect of bariatric surgery on male reproductive function.

ELIGIBILITY:
Inclusion Criteria:

* Meet the surgical indications according to the Chinese Guidelines for Surgical Treatment of Obesity and Type 2 Diabetes (2019 Edition).
* 20 years old< patient<60 years old.
* Male

Exclusion Criteria:

* Incapacity of giving an informed consent.
* Drug and / or alcohol abuse.
* Scrotal injury and previous scrotal surgery.
* Use of phosphodiesterase-5 inhibitors.
* Mental illnesses that may affect compliance with clinical research, including dementia, active psychosis, major depression, or attempted suicide.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: bariatric surgery male candidate
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Semen quality assessment | 3 months after surgery
  Semen quality assessment based the following indicators, including the time of liquefaction, semen PH, semen volume, sperm numbers, sperm vitality, sperm motility, sperm morphology, concentration of zinc in seminal plasma, concentration of fructose in seminal plasma, concentration of neutral α-glucosidase in seminal plasma, concentration of seminal elastase.The corresponding detection method is based on WHO laboratory manual for the Examination and processing of human semen(FIFTH EDITION).

SECONDARY OUTCOMES:
Concentration of interleukin in plasma | baseline- 3 months -6 months-12 months-2 years-3years
  interleukin 6, interleukin 8, tumor necrosis factor-α
Change of body mass index Body constant | baseline- 3 months -6 months-12 months-2 years-3years
  Body mass index=weight(kg)/ height(m2)
Changes of Vitamins | baseline- 3 months -6 months-12 months-2 years-3years
  Vitamin A, Vitamin B1, Vitamin B2, Vitamin B9, Vitamin B12, Vitamin C, Vitamin D. Folic acid; Vitamin E.
Changes of micronutrient | baseline- 3 months -6 months-12 months-2 years-3years
  Copper, Zinc, Calcium, Magnesium, Iron, Selenium.
Changes of sex hormone | baseline- 3 months -6 months-12 months-2 years-3years
  Testosterone, estradiol, luteinizing hormone, prolactin, follicle stimulating hormone, progesterone.
Changes of Blood lipids | baseline- 3 months -6 months-12 months-2 years-3years
  High density lipoprotein; low density lipoprotein; cholesterol; triglyceride
Oral glucose tolerance test | baseline- 3 months -6 months-12 months-2 years-3years
  glucose-0,30,120min; C peptide-0,30,120min; insulin-0,30,120min.
Changes in International Index of Erectile Function-5 scale scores | baseline- 3 months -6 months-12 months-2 years-3years
  minimum point 0, maximum points 25, (≥22 points are normal, 17-21 mild Erectile dysfunction, 12-16 moderateErectile dysfunction, 8-11 moderate Erectile dysfunction, <7 severe Erectile dysfunction)
Changes Waist to hip ratio | baseline- 3 months -6 months-12 months-2 years-3years
  Waist to hip ratio(WHR)=waist(cm)/hip(cm)
Semen quality assessment | baseline-6 months-12 months-2 years-3years
  Semen quality assessment based the following indicators, including the time of liquefaction, semen PH, semen volume, sperm numbers, sperm vitality, sperm motility, sperm morphology, concentration of zinc in seminal plasma, concentration of fructose in seminal plasma, concentration of neutral α-glucosidase in seminal plasma, concentration of seminal elastase.The corresponding detection method is based on WHO laboratory manual for the Examination and processing of human semen(FIFTH EDITION).

CONTACTS AND LOCATIONS:
Overall Officials: Shaihong Zhu, M.D., Principal Investigator — Central South University Third Xiangya Hospital
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao X, Li P, Wang G, Li W, Song Z, Zhu S, Zhu L. Effect of laparoscopic sleeve gastrectomy on male reproductive function in Chinese men with obesity: a prospective cohort study. Int J Surg. 2024 Jun 1;110(6):3373-3381. doi: 10.1097/JS9.0000000000001328. PMID 38477110